CLINICAL TRIAL: NCT00831948
Title: Identification of Large-Scale Mutations of POLG Gene by QMPSF in Patients With Mitochondrial DNA Instability.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Centre Hospitalier Universitaire de Nice, Département de la Recherche Clinique et de l'Innovation
Other Study IDs: 08-CIR-02- Dr ROUZIER
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Mitochondrial Diseases; Diagnosis; DNA Mutations
MeSH Terms: conditions — Mitochondrial Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitochondrial disease: Patients already diagnosed for mitochondrial pathology without mtDNA mutations yet detected by current diagnostic techniques
  Interventions: Genetic: mitochondrial DNA mutations diagnosis

INTERVENTIONS:
Genetic: mitochondrial DNA mutations diagnosis — Identification of large-scale mutations of POLG gene by QMPSF in patients with mitochondrial DNA instability.

SUMMARY:
Mitochondrial diseases are a heterogeneous group caused by genetic defects in mitochondrial DNA or in nuclear genes. POLG is the most frequently involved gene in mtDNA instability diseases resulting in mtDNA multiple deletion and/or depletion. It encodes the DNA polymerase gamma (POLγ), the only known DNA polymerase found in mammalian mitochondria. Mutations in POLG could explain 45% of familial progressive external ophtalmoplegia associated with multiple mtDNA deletions. However, in more than 70%, the analysis of the genes involved in mtDNA instability remains unsuccessful.

To date, these genes are screened by sequencing methods that are not able to detect large-scale rearrangements. In order to detect possible large-scale rearrangements, the investigators propose to develop a new assay based on QMPSF (Quantitative Multiplex PCR of Short fluorescent Fragments) able to detect exon deletions and duplications. the investigators propose to screen the POLG gene by QMPSF in at least twenty patients with either no mutation or only one mutation detected in POLG and no mutation in other genes such as TWINKLE and ANT1.

This study would allow the investigators to know if large-scale rearrangements occur in the POLG gene and to estimate their frequency in patients with mtDNA instability. These data are important to know if the sequencing analysis of POLG should be completed by the screening for partial deletions and duplications to ensure an accurate molecular diagnosis of these syndromes. Moreover, this method could be extended to ANT1 and TWINKLE genes.

ELIGIBILITY:
Inclusion Criteria:

* Patients already diagnosed for mitochondrial pathology without mtDNA mutations yet detected by current diagnostic techniques

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients already diagnosed for mitochondrial pathology without mtDNA mutations yet detected by current diagnostic techniques
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-12

PRIMARY OUTCOMES:
Improving the diagnosis of mitochondrial pathology | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Cécile ROUZIER, MD, Principal Investigator — Centre Hospitalier Universitaire
Locations (1):
- Centre Hospitalier Universitaire de Nice- Hôpital ARCHET 2 -Laboratoire de Génétique Médicale, Nice, France